CLINICAL TRIAL: NCT01115465
Title: Real-time Observation of Safety and Effectiveness in the Treatment of Female Stress Urinary Incontinence
Brief Title: Study of Macroplastique Safety and Effectiveness in the Treatment of Female Stress Urinary Incontinence
Acronym: ROSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uroplasty, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPQ092006
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; silicone elastomer
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macroplastique (Other): Macroplastique will be used for the treatment in an open-label, five year, post-market study
  Interventions: Device: Macroplastique

INTERVENTIONS:
Device: Macroplastique — Macroplastique is an injectable soft-tissue bulking agent used to treat stress urinary incontinence (SUI) primarily due to intrinsic sphincter deficiency (ISD).
  Other Names: polydimethylsiloxane; PDMS

SUMMARY:
The ROSE Registry will determine the long-term safety and effectiveness of Macroplastique in the treatment of female stress urinary incontinence (SUI) due to intrinsic sphincter deficiency (ISD).

DETAILED DESCRIPTION:
The Rose Registry is a five-year post-market study of the safety and effectiveness of Macroplastique in the treatment of female stress urinary incontinence due to intrinsic sphincter deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed written informed consent
* Subject is a female at least 18 years of age
* Subject has been diagnosed with SUI primarily due to intrinsic sphincter deficiency (ISD)
* Subject understands all study requirements including five year follow-up schedule
* Subject is psychologically stable and suitable for intervention as determined by the Investigator

Exclusion Criteria:

* Subject has an acute urogenital tract inflammation or infection
* Subject is pregnant or intends to become pregnant within one year
* Subject has had a sling placement within 12 weeks
* Subject has had a bulking agent treatment within 12 weeks
* Subject has a bladder neck or urethral stricture, gross utero-vaginal prolapse, untreated detrusor instability or hyperreflexia, neuropathic bladder, or overflow incontinence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
To describe the incidence of additional or alternative treatment for stress urinary incontinence due to ISD following up to two Macroplastique treatments over a 5 year period. | 5-years
  To describe the incidence of additional or alternative treatments

SECONDARY OUTCOMES:
To describe the incidence of genitourinary and treatment related adverse events, including transient symptoms associated with the injection procedure. | 5-years
  To describe the incidence of genitourinary and treatment related adverse events

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Kaiser Permanente Southern California-Irvine Medical Center, Irvine, California
  - Univeristy of California- Irvine, Orange, California
  - The University of California- of San Diego, San Diego, California
  - Urology Associates, PC, Englewood, Colorado
  - Specialists in Urology, Naples, Florida
  - The Florida Bladder Institute, Naples, Florida
  - Northwestern University Prentice Women's Hospital, Chicago, Illinois
  - Deaconess Clinic, Newburgh, Indiana
  - The University of Michigan Health Center, Ann Arbor, Michigan
  - Mercy Heatlh Partners at the Lakes, Muskegon, Michigan
  - Western New York Urology, Cheektowaga, New York
  - Western Carolina Women's Specialty Center, Asheville, North Carolina
  - Carolina Urology Partners, Gastonia, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Southern Urogynecology, Columbia, South Carolina
  - Urology of Virginia, Virginia Beach, Virginia
  - Athena Urology, Issaquah, Washington

IPD SHARING:
Plan to Share IPD: No